CLINICAL TRIAL: NCT06278740
Title: Investigation of Upper Extremity Pathologies and Associated Factors in Patients With Spinal Cord Injuries
Brief Title: Upper Extremity Pathologies in Spinal Cord Injuries
Status: Completed | Type: Observational
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Mahmut Sami Doğanlar, Medical Doctor, Afyonkarahisar Health Sciences University
Other Study IDs: SCIUSG24
Record Dates: First submitted 2024-02-19; First posted 2024-02-26 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2024-08

CONDITIONS: Spinal Cord Injuries; Upper Extremity Problem; Musculoskeletal Pain
MeSH Terms: conditions — Spinal Cord Injuries; Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SCI with Manual Wheelchair Usage: Patients with spinal cord injuries who use manual wheelchairs
  Interventions: Diagnostic Test: Musculoskeletal Ultrasound
- SCI without Manual Wheelchair Usage: Patients with spinal cord injuries who do not use manual wheelchairs
  Interventions: Diagnostic Test: Musculoskeletal Ultrasound

INTERVENTIONS:
Diagnostic Test: Musculoskeletal Ultrasound — Upper extremity pathologies of participants with ultrasound

SUMMARY:
This study aims to determine the relationship between upper extremity pathologies and demographic data, duration of manual wheelchair use, duration of injury, physical examination and musculoskeletal ultrasound measurements in patients with spinal cord injuries.

DETAILED DESCRIPTION:
Spinal cord injury is a neurological condition that can result from traumatic or non-traumatic causes, leading to motor, sensory and autonomic dysfunctions. Following a spinal cord injury, the upper extremity becomes increasingly used for mobility, weight-bearing, and transfer activities, making functionality crucial in daily life. Wheelchairs, commonly used by individuals with spinal cord injuries for daily activities, can lead to injuries and pain or degeneration in the upper extremities due to repetitive transfer activities. As a result, individuals with spinal cord injuries are at high risk for shoulder, elbow, wrist and hand injuries. Neuromuscular ultrasound (NMUS) has become increasingly important in clinical use in the evaluation of peripheral nerves and muscles in patients with spinal cord injuries in recent years, due to the advantages of ultrasonography such as providing dynamic and real-time evaluation, not containing radiation, and being painless.

This study aims to determine the relationship between upper extremity pathologies and demographic data, duration of manual wheelchair use, duration of injury, physical examination and musculoskeletal ultrasound measurements in patients with spinal cord injuries.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have experienced spinal cord injury, can comply with two-stage verbal commands, voluntarily agree to participate in the study and are medically stable.

Exclusion Criteria:

* Tetraplegia
* A significant comorbid condition such as severe heart disease and uncontrolled hypertension.
* Cognitive dysfunction
* Active infection
* Malignancy
* History of trauma to the upper extremity
* Brachial plexus and peripheral nerve injury
* History of surgery on the upper extremity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Spinal cord injuries who use manual wheelchairs and spinal cord injuries who do not use manual wheelchairs, aged between 18-65 years who applied to our clinic will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2024-08-05 (Actual); Primary Completion 2025-10-04 (Actual); Study Completion 2025-10-04 (Actual)

PRIMARY OUTCOMES:
Comparison of US findings among participants | 1 day (a single point in time)
  Ultrasonographic evaluation of upper extremity shoulder, elbow and wrist pathologies and examination of their relationship with clinical parameters.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | 1 day (a single point in time)
  Pain intensity was measured with visual analogue scale for pain (0-10 mm; 0 means no pain, 10 means severe pain) which is used to measure musculoskeletal pain with very good reliability and validity.
The Physical Examination of the Shoulder Scale (PESS) | 1 day (a single point in time)
  Includes 10 specific shoulder examination methods (Neer test, Hawkins test, Painful arc test, Supraspinatus test, Speed test, Yergason's test, O'brien test, Gerber's lift-off test, Horizontal adduction test, 0-degree abduction test). For each test, if there is no pain, 0 points are given; if there is suspected pain, 1 point is given; if there is obvious pain described during the test, 2 points are given. The maximum score for a single shoulder is 20 points.
The Quick Disability of the Arm, Shoulder, and Hand (Quick DASH) | 1 day (a single point in time)
  Quick DASH is a rapid, practical, and frequently used scale that allows the evaluation of the functional and symptomatic status of patients with upper extremity problems. The questionnaire consists of 11 questions, with 5 options provided for each question. A higher score indicates more activity limitation and greater difficulty.
American Spinal Injury Association (ASIA) Impairment Scale | 1 day (a single point in time)
  ASIA assessment consists of two parts: motor and sensory. Motor assessment involves testing the strength of ten key muscles on each side of the body in the supine position (ranging from 0 = no contraction to 5 = normal resistance). The maximum score for the upper extremities and lower extremities is 50. Sensory evaluation includes testing pinprick and light touch sensation. Pinprick and light touch sensations are scored separately for each dermatome on a 3-point scale (0, 1, and 2). Total highest score is 224, higher score indicates better.
The Spinal Cord Independence Measure (SCIM-III) | 1 day (a single point in time)
  Reliable tool for measuring the level of independence following spinal cord injury (SCI). The total score ranges from 0 to 100 and comprises sub-items such as Personal Care (0-20), Respiration and Sphincter Management (0-40), and Mobility (0-40). Lower scores indicate decreased levels of independence.

CONTACTS AND LOCATIONS:
Overall Officials: Mahmut Sami DOĞANLAR, MD, Principal Investigator — Afyonkarahisar Health Sciences University; Nuran EYVAZ, MD, Principal Investigator — Afyonkarahisar Health Sciences University
Locations (2):
- Turkey (Türkiye) (2):
  - Afyonkarahisar, Afyonkarahisar, Afyonkarahisar
  - Afyonkarahisar Health Sciences University, Afyonkarahisar, Afyonkarahisar

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ata AM, Mete Civelek G, Kara O. Relationship Between Manual Wheelchair Using Skills and Upper Limb Musculoskeletal Disorders in Patients With Spinal Cord Injury: A Musculoskeletal Ultrasonography Study. Am J Phys Med Rehabil. 2023 Nov 1;102(11):959-964. doi: 10.1097/PHM.0000000000002296. Epub 2023 May 23. PMID 37256679
- [Background] Collinger JL, Fullerton B, Impink BG, Koontz AM, Boninger ML. Validation of grayscale-based quantitative ultrasound in manual wheelchair users: relationship to established clinical measures of shoulder pathology. Am J Phys Med Rehabil. 2010 May;89(5):390-400. doi: 10.1097/PHM.0b013e3181d8a238. PMID 20407304
- [Background] Vives Alvarado JR, Felix ER, Gater DR Jr. Upper Extremity Overuse Injuries and Obesity After Spinal Cord Injury. Top Spinal Cord Inj Rehabil. 2021;27(1):68-74. doi: 10.46292/sci20-00061. PMID 33814884
- See also: Relationship Between Manual Wheelchair Using Skills and Upper Limb Musculoskeletal Disorders in Patients With Spinal Cord Injury: A Musculoskeletal Ultrasonography Study — https://pubmed.ncbi.nlm.nih.gov/37256679/
- See also: Validation of Greyscale-Based Quantitative Ultrasound in Manual Wheelchair Users — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC2859462/
- See also: Upper Extremity Overuse Injuries and Obesity After Spinal Cord Injury — https://pubmed.ncbi.nlm.nih.gov/33814884/